CLINICAL TRIAL: NCT04596670
Title: 68Ga-ICAM-1pep PET/CT Imaging of Tumor Responses to Radiotherapy in Cancer Patients
Brief Title: 68Ga-ICAM-1pep PET/CT in Cancer Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University Health Science Center (Other)
Responsible Party: Principal Investigator, Hua Zhu, Principal Investigator and Vice Director, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020KT112
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cancer
Keywords: PET/CT; Radiotherapy; ICAM-1; 68Ga labeling
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-ICAM1-1pep PET/CT in cancer patients before radiotherapy (Experimental): Cancer patients who have not undergone radiotherapy will be injected with 2.96 MBq/kg body weight of 68Ga-ICAM-1pep in one dose intravenously and then undergo PET/CT scan 1 h later.
  Interventions:
  Drug: 68Ga-ICAM-1pep Device: PET/CT
  Interventions: Drug: 68Ga-ICAM-1pep
- 68Ga-ICAM1-1pep PET/CT in cancer patients after radiotherapy (Experimental): Cancer patients post-radiotherapy will be injected with 2.96 MBq/kg body weight of 68Ga-ICAM-1pep in one dose intravenously and then undergo PET/CT scan 1 h later.
  Interventions:
  Drug: 68Ga-ICAM-1pep Device: PET/CT
  Interventions: Drug: 68Ga-ICAM-1pep

INTERVENTIONS:
Drug: 68Ga-ICAM-1pep — 68Ga-ICAM-1pep PET/CT: after intravenous injection of 2.96 MBq/kg body weight of quality-controlled 68Ga-ICAM-1pep, a Siemens Biograph PET/CT scan will be applied within 1 h, and the scan range will be from the top of the head to 1/3 of the upper thigh.
  Other Names: 68Ga-CD54pep

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the clinical predictive value of 68Ga-ICAM-1pep in metastatic cancer patients receiving radiotherapy. A single dose of 2.96 MBq/kg body weight of 68Ga-ICAM-1pep will be injected intravenously. The visual and semiquantitative methods will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
Radiotherapy has a systemic inhibitory effect on non-irradiated lesions (abscopal effect) in addition to local antitumor effects, and currently no biomarkers are used for the prediction of the abscopal effect of radiotherapy in standard clinical practice. Our recent preclinical studies identified ICAM-1 as a potential predictive biomarker for the radiotherapy-induced abscopal effect. In this clinical trial, we aim to investigate whether the ICAM-1-targeting radiotracer 68Ga-ICAM-1pep could be used for PET imaging of tumor responses to radiotherapy in cancer patients. PET/CT imaging of 68Ga-ICAM-1pep will be performed in patients before and after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. ECOG score 0 or 1 point;
3. Patients with suspected or confirmed lung cancer, esophagus cancer, cervical cancer or other cancers who are suggested by the clinicians to conduct PET/CT imaging for tumor diagnosis or staging.

Exclusion Criteria:

1. Pregnant or nursing;
2. Severe hepatic or renal dysfunction;
3. Low WBC (less than 3 x 10^9/L);
4. Unable to comply with the PET/CT imaging procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitate the standardized uptake values (SUVs) of 68Ga-ICAM-1pep at baseline. | At baseline
  Perform PET/CT imaging using 68Ga-ICAM-1pep before radiotherapy.The semiquantitative analysis will be performed by the same nuclear medicine physician for all cases, and the standardized uptake values (SUVs) of 68Ga-ICAM-1pep in the tumor lesions will be measured.
Characterize changes in the standardized uptake values (SUVs) of 68Ga-ICAM-1pep during radiotherapy. | 3 to 4 weeks after beginning of radiotherapy
  Perform PET/CT imaging using 68Ga-ICAM-1pep after radiotherapy. The semiquantitative analysis will be performed by the same nuclear medicine physician for all cases, and the standardized uptake values (SUVs) of 68Ga-ICAM-1pep in the tumor lesions will be measured. The SUVs of 68Ga-ICAM-1pep in the tumor lesions after radiotherapy will be compared with that at the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yang, Ph.D, Study Chair — Peking University Cancer Hospital & Institute; Hua Zhu, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Zhang T, Wang Y, Lu D, Du J, Feng X, Zhou H, Liu N, Zhu H, Qin S, Liu C, Gao X, Yang Z, Liu Z. ICAM-1 orchestrates the abscopal effect of tumor radiotherapy. Proc Natl Acad Sci U S A. 2021 Apr 6;118(14):e2010333118. doi: 10.1073/pnas.2010333118. PMID 33785590